CLINICAL TRIAL: NCT04359238
Title: activeDCM - Interventional Clinical Trial of Individualized Activity and Exercise Programs to Improve Outcome in Dilated Cardiomyopathy Guided by Longitudinal Biosensing With Apple Watch
Acronym: ACTIVE-DCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Apple Inc. (Industry); The German Heart Foundation (Other); Informatics for Life (Unknown); e-Cardiology (Unknown); German Cardiac Society (Other); Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Principal Investigator, Benjamin Meder, Prof. Dr. med., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTIVE-DCM
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cardiomyopathy, Dilated; Heart Failure
Keywords: Exercise; SmartWatch; Wearables; Digital Health; Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group with motivation messages (Active Comparator): There are 100 patients in the intervention group with automated or observer initiated motivation messages. They receive an individualized training program with regular notifications about their training status via their SmartWatch.
  Interventions: Behavioral: Individualized excercise
- Intervention group without motivation messages (Active Comparator): There are 100 patients in the intervention group without automated or observer initiated motivation messages. They receive an individualized training program without regular notifications about their training status via their SmartWatch.
  Interventions: Behavioral: Individualized excercise
- Control group (No Intervention): 100 patients are in the control group without an individualized training program.

INTERVENTIONS:
Behavioral: Individualized excercise — The participants in the intervention group carry out regularly endurance and strength exercises.
  Arms: Intervention group with motivation messages; Intervention group without motivation messages

SUMMARY:
The influence of an individualized sports program on dilated cardiomyopathy patients will be investigated in a randomized, prospective intervention study. 300 patients with dilated cardiomyopathy are included and examined over a period of 13 months. All participants will receive an Apple Watch, which serves for monitoring of activity and symptoms.The primary endpoint of the study is the change in maximum oxygen intake. In addition, the changes in well-being, objective parameters of cardiac function and the subject's compliance to his excercise program are of interest as secondary endpoints and for further exploratory research. In addition, the safety of a personalized sports program is evaluated. Molecules circulating in the blood (including proteins, RNA) are beeing measured at the beginning and in the course of the training program in order to be able to derive a connection between the training and the changed cardiovascular function. A gene analysis will be carried out, which serves to identify the genetic requirements of protective excercise.

DETAILED DESCRIPTION:
The recruited subjects (n = 300) receive routine medical care on the day of randomization in our outpatient clinic. Furthermore, an additional blood sample is taken (further blood samples are taken on month 6 and month 12), which contain 9 ml EDTA (for DNA analysis, e.g. whole genome sequencing), 5 ml of PaxGene (for RNA analysis), 7.5 ml of plasma (for example for metabolite and RNA analysis) and 7.5 ml of serum (for example for metabolite and RNA analysis). A detailed medical history is taken during the basic examination. This is followed by detailed physical examination and diagnostics. A routine blood sample is taken to determine the values of electrolytes, NT-ProBNP, hsTnT, creatinine, urea and the blood count. Finally, the patients answer a questionnaire on Quality of Life (MHLFQ: The Minnesota Living with Heart Failure Questionnaire) and Depression (PHQ9).

Two thirds of the patients (n = 200; intervention groups) will regularly participate in an individually designed sports program for a period of 12 months. One third of the participants (n = 100; control group) will not participate in a sports program. As a SmartWatch is required for the study. SmartWatches will be made available to all subjects on the day of recruitment. These are Apple Watches (Series 4), which are provided by Apple Inc. On the Apple Watch, participants have access to an app, that was especially developed by us for the study. This app collects important information about the physical activity and symptoms of the patient (including pulse rate, duration of training, the number of floors, number of steps and ECGs). The Apple Watch is also used to send participants of the intervention group regular notifications about their training status and to remind them of their training.

The participants present themselves 4-6 weeks after recruitment in the department of sports medicine to perform a spiroergometry and a sports medical evaluation. A personalized sports program (depending on the severity of the disease) is created for the subjects of the intervention groups, which consists of strength and endurance training. The sports program will be carried out over a period of 12 months.

All subjects in the intervention groups receive follow-up visits on month 3, month 6, month 9 and month 12. The sports program can be adapted on these dates. The subjects who did not receive a personalized training program presente themselves for the follow-up examination on month 6 and month 12. Unwanted events during the training (including syncope, ICD therapy, injuries) are documented during the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-ischemic, dilated cardiomyopathy (DCM)
* EF ≤ 45%
* NYHA I-III
* Age 18 to 65 years
* The patient understood the study concept and the declaration of consent and signed and dated the declaration of consent

Exclusion Criteria:

* Physical disability that is not compatible with exercise in the study
* Orthopedic diseases such as osteoarthritis or changes in the spine that lead to restrictions that are not compatible with exercise in the study
* Syncope within the past 3 months
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum oxygen uptake (VO2max) | 12 months
  Change in maximum oxygen uptake (VO2max) from baseline to 12 months follow-up

SECONDARY OUTCOMES:
Quality of life (Patient Reported Outcome) | 12 months
  Change in quality of life

OTHER OUTCOMES:
Cardiac biomarkers | 12 months
  Change in Troponin und NTproBNP
Cardiac function | 12 months
  Change in systolic and diastolic cardiac function
Arrhythmias | 12 months
  Change in frequency of arrhythmias
Heart failure | 12 months
  Change in frequency of hospitalization and NYHA class
Compliance | 12 months
  Change in compliance concerning excercise program

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Meder, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- Department III of Internal Medicine, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided